CLINICAL TRIAL: NCT06978426
Title: Evaluation of Grip Strength Asymmetry Index in Professional E-Sports Athletes as a Predictive Measure for Wrist Pain
Brief Title: Hand-Held Dynamometer Assessment: E-Sports Grip-Asymmetry Index as a Predictor of Wrist Pain
Status: Recruiting | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy, Ahram Canadian University
Other Study IDs: AlHayah-1001
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Wrist Injuries
MeSH Terms: conditions — Wrist Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain Group: Professional e-sports athletes reporting wrist pain ≥3/10 on VAS during play
  Interventions: Other: Pain Group
- No-Pain Group: Professional e-sports athletes reporting minimal to no wrist pain (<3/10 on VAS during play)
  Interventions: Other: No-Pain Group

INTERVENTIONS:
Other: Pain Group — Professional e-sports athletes who report wrist pain rated at 3 or higher on a 10-point Visual Analog Scale during gaming activities. These participants play video games professionally for at least 35 hours per week, are between 18-30 years old, and have no history of neurologic or rheumatic disease.
  Groups: Pain Group
Other: No-Pain Group — Professional e-sports athletes who report minimal to no wrist pain (less than 3 on a 10-point Visual Analog Scale) during gaming activities. These participants play video games professionally for at least 35 hours per week, are between 18-30 years old, and have no history of neurologic or rheumatic disease.
  Groups: No-Pain Group

SUMMARY:
This cross-sectional study investigates whether a simple Grip-Asymmetry Index (GAI) can predict self-reported wrist pain in professional e-sports athletes. Professional gamers (aged 18-30) who play at least 35 hours per week will be assessed using a Jamar dynamometer to measure maximal grip force in both hands. The study will compare GAI between two groups: those with wrist pain (≥3/10 on Visual Analog Scale during play) and those without pain. A GAI cutoff value for predicting wrist pain risk will be established through ROC analysis, with additional factors such as gaming hours, BMI, and sex incorporated into a multivariable logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Professional e-sports athletes (receiving compensation for gaming activities)
* Age between 18 and 30 years
* Gaming for at least 35 hours per week
* For Pain Group: Reports wrist pain rated ≥3/10 on VAS during gaming activities
* For No-Pain Group: Reports minimal to no wrist pain (<3/10 on VAS) during gaming activities

Exclusion Criteria:

* History of neurologic disease
* History of rheumatic disease
* Previous wrist surgery
* Recent wrist trauma (within 3 months)
* Use of pain medication within 24 hours of assessment
* Inability to perform grip strength testing

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Professional e-sports athletes between 18-30 years old who compete in organized video gaming competitions and receive compensation for their gaming activities. Participants will be recruited from professional e-sports teams, gaming organizations, and competitive gaming events in the region. The study population will include individuals who play competitive video games for at least 35 hours per week using standard computer peripherals (mouse and keyboard). Both male and female athletes will be eligible, and efforts will be made to recruit a representative sample across different gaming genres (FPS, MOBA, RTS, etc.) and competitive levels.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Grip-Asymmetry Index (GAI) | Measured once at study enrollment
  The Grip-Asymmetry Index is calculated as (Dominant hand grip strength - Non-dominant hand grip strength) / Dominant hand grip strength × 100%. Grip strength is measured in kilograms using a calibrated Jamar hand-held dynamometer following standardized testing protocols. Higher GAI values indicate greater asymmetry between dominant and non-dominant hands.

SECONDARY OUTCOMES:
Maximal grip force in dominant hand | Measured once at study enrollment
  Maximum grip strength measured in kilograms using a calibrated Jamar hand-held dynamometer following standardized testing protocols
Maximal grip force in non-dominant hand | Measured once at study enrollment
  Maximum grip strength measured in kilograms using a calibrated Jamar hand-held dynamometer following standardized testing protocols
Wrist pain intensity during gaming | Assessed at study enrollment, reflecting current pain experience during gaming activities
  Self-reported wrist pain measured using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable) during typical gaming sessions
Weekly gaming hours | Assessed at study enrollment, reflecting average from the past month
  Self-reported average number of hours spent gaming per week

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No